CLINICAL TRIAL: NCT05741567
Title: Transobturator Cystocele Repair by Vaginal Plastron
Brief Title: Transobturator Repair by Vaginal Plastron
Acronym: CYSPTO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5083; 69HCL22_1180 (Other: HCL)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Anterior Prolapse Surgery Using the Transobturator Repair by Vaginal Plastron
Keywords: anterior prolapse; transobturator repair; vaginal plastron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- transobturator cystocele repair by vaginal plastron: patients who underwent surgery using the transobturator repair by vaginal plastron for correction of anterior prolapse
  Interventions: Procedure: correction of anterior prolapse

INTERVENTIONS:
Procedure: correction of anterior prolapse — percentage of failed prolapse correction

SUMMARY:
The autologous vaginal route consists of repairing the genital prolapse through the vagina using the patient's tissues without a prosthesis. Vaginal prostheses are actually currently prohibited in France [1, 2].

The autologous vaginal route is the quickest surgery and it can be done under spinal anesthesia, which constitutes arguments for offering it to elderly and fragile patients. The autologous vaginal approach gives functional and subjective results similar to promontofixation [2].

There are many surgical techniques that make it difficult to assess the recurrence rate in the literature. Autologous vaginal surgery provides a good degree of satisfaction for patients despite the risk of recurrence [3].

We propose to describe the results of the transobturator cystocele repair by vaginal plastron, a technique which seems reproducible and effective to us.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* patient who underwent surgery using the transobturator repair by vaginal plastron for correction of anterior prolapse requiring surgical correction of stage equal to or greater than II in the POP-Q classification
* intervention between September 2020 and October 2022
* person having expressed his non-opposition

Exclusion Criteria:

* inability to understand the information given
* person deprived of liberty
* person under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study covers all patients who underwent surgery using the transobturator repair by vaginal plastron for correction of anterior prolapse between September 2020 and October 2022.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
failed prolapse correction | at 1 month after surgery
  percentage of failed prolapse correction

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Lyon, BRON, France